CLINICAL TRIAL: NCT06061562
Title: Down Syndrome, Physical Activity and Sleep Apnea
Acronym: TAPAS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0146
Record Dates: First submitted 2023-06-15; First posted 2023-09-29 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Down Syndrome
Keywords: Down syndrome; sleep disorders; Apnea; physical activity; neurocognition; autonomic nervous system
MeSH Terms: conditions — Down Syndrome; Sleep Wake Disorders; Apnea; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — blood samples to analyze inflammatory profile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DS group: A cohort of participants (child, teenager, or adult), with or without sleep disorders

SUMMARY:
To realize a sleep phenotyping in a population with Down syndrome, its determinants, and the consequences of these disorders, with a specific focus on sleep apnea syndrome.

DETAILED DESCRIPTION:
Sleep disorders are widely observed in the Down's syndrome population, due to a number of risk factors, and can become established in early childhood. Diagnosis of sleep disorders in Down's syndrome is difficult and often delayed, which can contribute to poor health in children with Down's syndrome. Phenotyping sleep characteristics in this Down Syndrome population will enable early identification of the consequences of these disorders, with a specific focus on sleep apnea syndrome, whose origin is multisystemic.

ELIGIBILITY:
Inclusion Criteria:

* Total autosomal trisomy caused by the presence of a third copy (partial or total) of chromosome 21

Exclusion Criteria:

* People with abnormal electrocardiographic tracings,
* Existence of heart failure or cardiovascular disease, as determined by any abnormalities in cardiovascular adaptations to exercise.
* Existence of a declared or uncontrolled progressive disease.
* pregnant or breast-feeding women.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Down syndrome is associated with numerous clinical expressions. The most frequent are deficits in cognitive development, autonomic nervous system dysfunctions, cardiovascular dysfunctions, and osteoarticular specificities. Taken together, these clinical features can lead to a sedentary and overweight lifestyle, directly responsible for the onset of early fatigue and effort limitation. Numerous co-morbidities are also reported, such as the presence of sleep apnea syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
phenotyping of sleep in a population with Down's syndrome, its determinants, and the consequences of these disorders, with a specific focus on sleep apnea syndrome, whose origin is multisystemic | Visite 2: 2 nights
  Diagnosis of Sleep Apnea Syndrome using calculation of apnea hypopnea index (AHI)>15 events/h

SECONDARY OUTCOMES:
Sleep-disordered breathing associated with dysautonomia | Visite 2: 1 night
  Polysomnography
Sleep-disordered breathing associated with dysautonomia | Visite 2: up to 3 nights
  Heart rate (beat per min) recording using a cardiofrequency meter to measure the RR interval (in milliseconds); measured over 3 nights max in an ecological environment
Sleep-disordered breathing associated with dysautonomia | Visite 2: up to 3 nights
  The variables used to assess the autonomic profile will be obtained by calculating LF and LF(low and high frequency in ms² and normalized units) spectral variations and the LF/HF ratio
Sleep-disordered breathing associated with specific abnormalities of the biological work-up | Visite 1: the morning before the physical activity
  Biological disturbances will be assessed by differences in thyroid function, and other biological variables (NFS, lipid and hormone levels, iron levels) in comparison with standards. This biological assessment is obtained by blood sampling.
Sleep-disordered breathing associated with a specific cranial structure | Day 0
  The existence of cranial anatomical variations, in particular anomalies specific to the oral sphere (modification of the gonia angle (in degrees), and prognatism (in cm)) will be investigated by cephalometry.
Sleep-disordered breathing associated with inadequate physical activity | Day 0 and visite 1
  Abnormalities in the physiological response to exercise (VO2 (in mL/kg/min) compared with the predicted value) will be investigated and linked to the level of physical activity measured by questionnaires (scores).
Sleep-disordered breathing associated with inadequate physical activity | From inclusion to last visit of the patient: up to 90 days
  Abnormalities in the physiological response to exercise (VO2 (in mL/kg/min) compared with the predicted value) will be investigated and linked to the level of physical activity measured by actimetry (min per day)
Sleep-disordered breathing associated with inadequate physical activity | Day 0 and visite 1: 1 time
  Abnormalities in the physiological response to exercise (VO2 (in mL/kg/min) compared with the predicted value) will be investigated and linked to the level of physical activity measured by anthropometric variables (Weight (kg)
Sleep-disordered breathing associated with inadequate physical activity | Day 0 and visite 1: 1 time
  Abnormalities in the physiological response to exercise (VO2 (in mL/kg/min) compared with the predicted value) will be investigated and linked to the level of physical activity measured by Height (m)
Sleep-disordered breathing associated with inadequate physical activity | Day 0 and visite 1: 1 time
  Abnormalities in the physiological response to exercise (VO2 (in mL/kg/min) compared with the predicted value) will be investigated and linked to the level of physical activity measured by BMI (kg/m²)
Sleep-disordered breathing associated with inadequate physical activity | Visite 1: up to 1 hour
  Abnormalities in the physiological response to exercise (VO2 (in mL/kg/min) compared with the predicted value) will be investigated and linked to the level of physical activity measured by determinants of physical fitness (measurement of strength (Newton)
Sleep-disordered breathing associated with inadequate physical activity | Visite 1: up to 1 hour
  Abnormalities in the physiological response to exercise (VO2 (in mL/kg/min) compared with the predicted value) will be investigated and linked to the level of physical activity measured by flexibility (cm)
Sleep-disordered breathing associated with inadequate physical activity | Visite 1: up to 1 hour
  Abnormalities in the physiological response to exercise (VO2 (in mL/kg/min) compared with the predicted value) will be investigated and linked to the level of physical activity measured by balance variables (seconds).
Sleep-disordered breathing associated with inadequate physical activity | Visite 1: up to 1 hour
  Effort response (% chronotropic response) will also be calculated to complete the autonomic profile.
Sleep-disordered breathing associated with specific neurobehavioral disorders | Day 0
  A neurobehavioral profile assessment will be carried out using several tests, in order to verify the possible impact of TdS on cognitive function:
  * Intelligence quotient (Wechsler scale), if not previously performed (score)
  * Stroop task (inhibitory control) (score)
  * Reaction time using a light device (seconds)
  * Ability to perform a double cognitive-motor task, (score)
  * BRIEF questionnaire (to explore executive function) (score)
  * ADHD rating scale (to explore signs of attention deficit/hyperactivity disorder). (score)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien BAILLIEUL, Principal Investigator — University Grenoble Hospital
Locations (1):
- Chu Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided